CLINICAL TRIAL: NCT03785392
Title: Out of Plane Approach for Interscalene Level Brachial Plexus Block to Avoid Phrenic Nerve Involvement - a Prospective Study
Brief Title: Out of Plane Approach for Interscalene
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary investigator left the Institution
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-0121
Record Dates: First submitted 2018-11-07; First posted 2018-12-24 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-10

CONDITIONS: Acute Pain; Brachial Plexus Block
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 Inplane (Active Comparator): Study with the technique Inplane group
  Interventions: Procedure: Group 1 In-plane
- Group 2 out of plane (Active Comparator): Study with the technique out of plane
  Interventions: Procedure: Group 2 out of plane

INTERVENTIONS:
Procedure: Group 1 In-plane — Group 1: Study will involve total of 15 patients with the procedure done in-plane. Before the block placement and after the block placement lung function will be measured.
  FEV1 (forced expiratory volume in 1 second ) and FVC ( forced vital Capacity ) values will be recorded. Block will be performed in plane and postprocedure lung function test will be repeated. New values of FEV1 and FVC will be obtained after the placement of the nerve block.
  Arms: Group 1 Inplane
Procedure: Group 2 out of plane — Group 2 study will adopt the out of plane technique and will involve a total of 15 patients in this group. We will do the procedure out of plane and will have lung function FEV1 and FVC measured bedside.FEV1 and FVC values will be recorded. Block will be performed out of plane and postprocedure lung function test will be measured. New values of FEV1 and FVC will be obtained
  Arms: Group 2 out of plane

SUMMARY:
Study aims to examine the influence of out of plane interscalene approach to a brachial plexus block on the effect of phrenic nerve blockade.

DETAILED DESCRIPTION:
Studies have proven that there is 100% blockade of the phrenic nerve with the in-plane approach to the interscalene brachial plexus block. The patient population with pulmonary comorbidities with poor reserve cannot afford to have a further deterioration of their pulmonary status due to phrenic nerve blockade. These patients are not ideal candidates for increased opiate therapy for intraoperative and post-surgical pain as well due to further depression of their respiratory function. To optimize their pain control as well as avoid any respiratory-related morbidity and mortality, it is ideal to develop a technique which can provide appropriate brachial plexus block at the interscalene level while completely avoiding any local anesthetic spread to the phrenic nerve.

The study aims to examine the influence of out of plane interscalene approach to a brachial plexus block on the effect of phrenic nerve blockade. Practitioner preference and institutional norms often influence the in plane approach for the above-mentioned block. The most common practice at our institution is the in plane approach to the brachial plexus block.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients(18-85 years old)
* Scheduled for elective shoulder surgery who would benefit from a preoperative interscalene approach to the brachial plexus block for intraoperative and postoperative pain relief.

Exclusion Criteria:

* Patients with any distorted anatomy for whom the block cannot be performed accurately, such as scars, surgical fixtures at the site, active infection, any open wound or drains at the site.
* Patients who request benzodiazepine anxiolytics such as midazolam for premedication before the procedure. Also patients who request narcotic medications as premedication before the procedure
* Non-English and Non-Spanish speaking patients
* Inadequate or failed blocks and inadvertently intrathecal or intravascular injection will be dropped from the study
* Incarcerated patients
* Expected heavy bleeding on multiple anticoagulants with markedly elevated PT ( Prothrombin time ), INR (International Normalized Ratio ), PTT ( Partial Thromboplastin Time ) levels and markedly reduced platelet counts

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2019-12-08 (Actual); Study Completion 2019-12-08 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume (FEV1) | The change in Forced Expiratory Volume in one second (FEV1) from Baseline to 15 minutes
  Forced Expiratory Volume in one second (FEV1) is measured in liters.

SECONDARY OUTCOMES:
Forced Vital Capacity (FVC) | The change in Forced Vital Capacity (FVC) from Baseline to 15 minutes
  Forced Vital Capacity (FVC) is measured in liters.

CONTACTS AND LOCATIONS:
Overall Officials: Ranganathan Govindaraj, MD, Principal Investigator — UTMB
Locations (2):
- United States (2):
  - UTMB, Galveston, Texas
  - UTMB, League City, Texas

IPD SHARING:
Plan to Share IPD: No